CLINICAL TRIAL: NCT05059613
Title: Study on Thalidomide With or Without Probiotics in Radioactive Oral Mucositis
Brief Title: Thalidomide With or Without Probiotics in Radioactive Oral Mucositis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Provincial Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: jcl2021-8
Record Dates: First submitted 2021-08-31; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Oral Mucositis; Quality of Life
MeSH Terms: conditions — Stomatitis | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- probiotics group (Experimental): Use thalidomide in combination with probiotics during radiotherapy and chemotherapy
  Interventions: Other: probiotics
- thalidomide group (No Intervention): Thalidomide is used only during radiotherapy and chemotherapy
- healthy control group (No Intervention): healthy control group

INTERVENTIONS:
Other: probiotics — one times a day during the whole treatment
  Arms: probiotics group

SUMMARY:
Study on the application of thalidomide with or without probiotics in radioactive oral mucositis

DETAILED DESCRIPTION:
Radiation oral mucositis is an acute mucous membrane reaction in patients undergoing radiotherapy of the head and neck. It can cause dose limitation and debilitating side effects. There is no accepted guideline that can significantly reduce its severity. In the mucosa, T and B cells of the immune system have location-specific phenotypes and functions that are influenced by the microbiome. These cells play a key role in maintaining immune homeostasis by inhibiting responses to harmless antigens and enhancing the integrity of intestinal mucosal barrier function. We designed a clinical study of thalidomide with or without probiotics in radioactive oral mucositis. The aim of this study was to determine whether regulation of intestinal flora can effectively reduce the severity of radiation-induced mucositis in patients undergoing radical radiation therapy. The researchers also investigated the effect of the intervention on patients' general well-being. The primary endpoint was the incidence of grade 3 mucositis in the radiotherapy oncology group. In 2021, an estimated 40 patients were enrolled in the study at Jiangxi Cancer Hospital in China.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky score ≥80 ,newly diagnosed NPC without distant metastasis, confirmed by pathology without any other malignant disease history ,no any other anti-cancer treatment for NPC previously ,received radiotherapy and chemotherapy at our Cancer Center

Exclusion Criteria:

* any immune system disease under high risk to antimicrobial agents such as Diabetes,infection disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-09-20 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of Radiation Therapy Oncology Group grade 3 mucositis | one month
  Radiation oral mucositis
the variaty of immune index | one month
  CD3,CD4,CD8
the variaty of immune index | one month
  Hemoglobin
the variaty of immune index | one month
  lymphocyte ratio

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, MD PHD, Principal Investigator — Jiangxi Provincial Cancer Hospital
Locations (1):
- Jiangxi Cancer Hospital, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: Undecided